CLINICAL TRIAL: NCT01517594
Title: Tolerability of Pentasa® Sachet in Patients With Ulcerative Colitis Under Conditions of Standard Practice in the Czech Republic
Brief Title: Tolerability of Pentasa Sachet in Patients With Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000026
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Confirmation of safety profile

ELIGIBILITY:
Inclusion Criteria:

* treatment of Ulcerative Colitis

Exclusion Criteria:

* hypersensitivity to mesalazine
* severe liver or renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
verify the safety profile: measured by number of AEs/SAEs | 12 months from patient recruitment

SECONDARY OUTCOMES:
dosage: evaluate dosage level | 12 months from patient recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (30):
- Czechia (30):
  - FN sv.Anna, Brno
  - Gastroenterologická ambulance, Brno
  - Hospital Milosrdných bratří, Brno
  - Hospital Břeclav, Břeclav
  - Nemocnice Cheb, Cheb
  - Nemocnice s poliklinikou Ráj, Fryštát
  - Gastroenterologická ambulance Hodonín, Hodonín
  - Hospital TGM Hodonín, Hodonín
  - FN, II. Interní klinika, Hradec Králové
  - Oblastní nemoncice Jičín, Jičín
  - Nemocnice Karlovy Vary, Karlovy Vary
  - Gastroenterologická ambulance Jezuitská, Litoměřice
  - Gastroenterologická ambulance Litoměřice, Litoměřice
  - GASTRO MED, s.r.o., Ostrava
  - Gastromedic s.r.o., Pardubice
  - 4. poliklinika Plzeň, Gastroenterologická ambulance, Pilsen
  - Fakultní poliklinika VFN, Prague
  - FN Motol, Prague
  - Iscare, Prague
  - Poliklinika - gastroenterologie, Prague
  - Poliklinika Clinicum - Interna, Prague
  - Sanatorium sv. Anny, Prague
  - Ústřední vojenská nemocnice, Prague
  - Hospital Prostějov, Prostějov
  - Poliklinika Mens, Přerov
  - Poliklinika - gastroenterologie Rychnov nad Kněžnou, Rychnov nad Kněžnou
  - Masarykova nemocnice,Interna, Ústí nad Labem
  - Nemocnice Valašské Meziříčí, Valašské Meziříčí
  - Vítkovická nemocnice, Vítkovice
  - Krajská nemocnice T.Bati, Zlín